CLINICAL TRIAL: NCT01674569
Title: A Phase 1 Open-label, Dose Escalation Clinical Trial to Evaluate the Safety and Preliminary Biologic Activity/Efficacy of the VEGFR/PDGFR Inhibitor X-82 Administered Per Os in Subjects With Neovascular Age-related Macular Degeneration (AMD)
Brief Title: Pilot Study of X-82 in Patients With Wet AMD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tyrogenex (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X82-OPH-102
Record Dates: First submitted 2012-08-23; First posted 2012-08-29 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Exudative Macular Degeneration
Keywords: VEGF; PDGF; AMD
MeSH Terms: conditions — Wet Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 50 mg X-82 oral alternate days (Experimental): 50 mg X-82 oral on alternate days with intravitreous ranibizumab (Lucentis) using predefined retreatment criteria for 24 weeks or until unacceptable toxicity develops
  Interventions: Drug: X-82 oral; Drug: ranibizumab (Lucentis)
- 50 mg X-82 oral QD (Experimental): 50 mg X-82 oral QD with intravitreous ranibizumab (Lucentis) therapy using predefined retreatment criteria.for 24 weeks or until unacceptable toxicity develops
  Interventions: Drug: X-82 oral; Drug: ranibizumab (Lucentis)
- 100 mg X-82 oral alternate days (Experimental): 100 mg X-82 oral on alternate days with intravitreous ranibizumab (Lucentis) using predefined retreatment criteria.for 24 weeks or until unacceptable toxicty develops
  Interventions: Drug: X-82 oral; Drug: ranibizumab (Lucentis)
- 100 mg X-82 oral QD (Experimental): 100 mg X-82 oral QD with intravitreous ranibizumab (Lucentis) using predefined retreatment criteria for 24 weeks or until unacceptable toxicity occurs
  Interventions: Drug: X-82 oral; Drug: ranibizumab (Lucentis)
- 200 mg X-82 oral QD (Experimental): 200 mg X-82 oral QD with intravitreous ranibizumab (Lucentis) therapy using predefined retreatment criteria for 24 weeks or until unacceptable toxicity occurs
  Interventions: Drug: X-82 oral; Drug: ranibizumab (Lucentis)
- 300 mg X-82 oral QD (Experimental): 300 mg X-82 oral QD with intravitreous ranibizumab (Lucentis) therapy using predefined retreatment criteria for 24 weeks or until unacceptable toxicity occurs.
  Interventions: Drug: X-82 oral; Drug: ranibizumab (Lucentis)

INTERVENTIONS:
Drug: X-82 oral — X-82 oral for 24 weeks or until unacceptable toxicity develops
Drug: ranibizumab (Lucentis) — Rescue treatment with intravitreal ranibizumab (Lucentis) as needed

SUMMARY:
The objective of this study is to evaluate the safety and preliminary biologic activity/efficacy of X-82 in patients with wet Age-related Macular Degeneration (AMD). Preliminary efficacy will be assessed by change from baseline in visual acuity, fluorescein leakage, retinal thickness and fibrosis, if detectable, based on fundus examination, fundus photography, fluorescein angiography and optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

1. Active choroidal neovascularization (CNV) associated with AMD, as evidenced on fluorescein angiography (FA) and OCT.
2. No previous treatment with anti-VEGF therapy or prior anti-VEGF therapy with evidence of response to treatment and the need for additional treatment.
3. Early Treatment Diabetic Retinopathy Study (ETDRS) BCVA 20/32 to 20/320 in the study eye(s).
4. Adequate bone marrow function.
5. PT within the institutional upper limit of normal.
6. Adequate hepatic function.
7. Adequate renal function; serum creatinine.
8. Ability to swallow oral medication.
9. Age ≥ 50 years.
10. Willing and able to provide written informed consent, comply with the investigational study protocol and return for all study visits.

Exclusion Criteria:

1. Previous treatment with photodynamic therapy (PDT) within 4 months of screening in the study eye.
2. CNV due to causes other than AMD.
3. Geographic atrophy involving the foveal center in the study eye.
4. Any retinal vascular disease or retinal degeneration other than AMD in the study eye.
5. In the opinion of the investigator, any significant disease in the study eye that could compromise best-corrected visual acuity.
6. Cataract surgery in the study eye within three months of screening.
7. Trabeculectomy or aqueous shunt or valve in the study eye.
8. Intraocular surgery in the study eye within three months of screening; Nd:YAG capsulotomy or laser iridotomy within 30 days of screening.
9. Inadequate pupillary dilation or significant media opacities in the study eye.
10. Use of any investigational agent or participation in any other clinical trial of an investigational agent or investigational therapy within thirty (30) days of baseline with the exception of subjects who are participating in the AREDS2 study.
11. Females of child bearing potential that are pregnant or not using medically acceptable contraception; males unwilling to take adequate contraceptive measures. Females that are breastfeeding are also excluded.
12. Serious allergy to or prior significant adverse reaction to fluorescein.
13. Undiagnosed acute illness first observed during screening or between screening and baseline, or severe concurrent medical conditions that, in the investigators judgment, represent a safety concern.
14. Severe cardiac disease, symptomatic congestive heart failure, unstable angina, acute coronary syndrome, myocardial infarction or coronary artery revascularization, or arterial thrombosis within 12 months of start of study drug, inadequately controlled hypertension, or ventricular tachyarrhythmias requiring ongoing treatment.
15. QTc ≥450 msec or subjects with a history of risk factors for Torsades de Pointes or other clinically significant ECG abnormalities as determined by the investigator.
16. Stroke or transient ischemic attack within 12 months of trial entry.
17. Clinically significant impaired renal or hepatic function.
18. Any major surgical procedure within one month of trial entry.
19. Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of X-82.
20. Receiving treatment with anti-coagulants other than 325 mg of aspirin per day.
21. Serious active infection, other serious medical condition or any other condition that would impair the ability of the subject to administer the investigational drug or to adhere to the study protocol requirements.
22. Presence of any condition which, in the judgment of the investigator, would prevent the subject from completing the study.
23. No herbal medications with the exception of bilberry are allowed within 7 days of start of study drug.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - New England Retina Associates, New London, Connecticut
  - Elman Retina Group, Baltimore, Maryland
  - Retina Research Institute of Texas, Abilene, Texas
  - Retina Consultants of Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jackson TL, Boyer D, Brown DM, Chaudhry N, Elman M, Liang C, O'Shaughnessy D, Parsons EC, Patel S, Slakter JS, Rosenfeld PJ. Oral Tyrosine Kinase Inhibitor for Neovascular Age-Related Macular Degeneration: A Phase 1 Dose-Escalation Study. JAMA Ophthalmol. 2017 Jul 1;135(7):761-767. doi: 10.1001/jamaophthalmol.2017.1571. PMID 28570723

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with wet age related macular degeneration were enrolled at 5 US retinal clinics between November 2012 and March 2015
Pre-assignment Details: 110 subjects were screened for entry into the study. 52 did not meet inclusion criteria, 19 declined to participate and 4 were excluded for other reasons
Groups:
- 50 mg X82 Alternate Days: Participants were assigned to 50 mg X-82 on alternate days for 24 weeks. After treatment discontinuation subjects were followed for an additional 4 weeks.
- 50 mg X82 QD: Participants were assigned to 50 mg X-82 QD for 24 weeks. After treatment discontinuation subjects were followed for an additional 4 weeks.
- 100 mg X82 on Alternate Days: Participants were assigned to 100 mg X-82 on alternate days for 24 weeks. After treatment discontinuation subjects were followed for an additional 4 weeks.
- 100 mg X82 QD: Participants were assigned to 100 mg X-82 QD for 24 weeks. After treatment discontinuation subjects were followed for an additional 4 weeks.
- 200 mg X82 QD: Participants were assigned to 200 mg X-82 QD for 24 weeks. After treatment discontinuation subjects were followed for an additional 4 weeks.
- 300 mg X82 QD: Participants were assigned to 300 mg X-82 QD for 24 weeks. After treatment discontinuation subjects were followed for an additional 4 weeks.
Period: Overall Study
Arm/Group | 50 mg X82 Alternate Days | 50 mg X82 QD | 100 mg X82 on Alternate Days | 100 mg X82 QD | 200 mg X82 QD | 300 mg X82 QD
Started | 3 | 8 | 4 | 10 | 7 | 3
Completed | 3 | 5 | 2 | 9 | 5 | 1
Not Completed | 0 | 3 | 2 | 1 | 2 | 2
Not completed — Adverse Event | 0 | 2 | 0 | 1 | 2 | 2
Not completed — Protocol Violation | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Escalation of X-82 and Ranibizumab Rescue: Groups of participants were assigned to 1 of 6 X-82 doses over 24weeks,with an additional 4 weeks for follow-up. The dose escalated from one level to the next in the absence of any dose-limiting toxicity (DLT) defined as a drug-related safety event during the first 2 weeks of treatment that was severe enough to require removal of the participant from the study.
  The escalating X82 oral dose regimens were 50 mg alternate days, 50 mg daily, 100 mg alternate days, 100mg daily, 200mg daily, and 300mg daily.
Arm/Group | Dose Escalation of X-82 and Ranibizumab Rescue
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35
Best corrected visual acuity [Mean (Standard Deviation); unit: Number of letters] | 62.4 (12.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Visual Acuity at 6 Months
Description: The best corrected visual acuity by the Early Treatment Diabetic Retinopathy Study (ETDRS) method was determined at baseline and at various times during the study. The ETDRS method records the number of letters of decreasing size on a chart that a subject can read from a defiend distance.
  During the study the ETDRS visual acuity was used to monitor the need for rescue therapy. The primary endpoint of the study was the change from baseline visual ETDRS visual acuity at 6 months. It was calculated by subtracting the baseline visual acuity from the visual acuity at 6 months for each individual subject. A positive change from baseline indicates improvement in visual acuity.
Time Frame: 6 months
Population: The mean and standard deviation was calculated for all subjects who completed 6 months of treatment with oral X82
Measure: Mean (Standard Deviation); unit: number of letters
Groups:
- All Completers: All subjects who successfully completed 6 months of treatment with oral X82
Arm/Group | All Completers
Number analyzed (Participants) | 25
number of letters | 3.8 (9.6)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for the duration of the study beginning at participant randomization and continuing till participant completion of the study. The participation of individual subjects in the study ranged from 1-7 months.
Description: Since the sample size for each dose group of X82 was limited, the frequency of adverse events are reported for all patients enrolled in the study.
Groups:
- Dose Escalation of X-82 and Ranibizumab Rescue: Groups of participants were assigned to 1 of 6 X-82 doses over 24 weeks,with an additional 4 weeks for follow-up. The dose escalated from one level to the next in the absence of any dose-limiting toxicity (DLT) defined as a drug-related safety event during the first 2 weeks of treatment that was severe enough to require removal of the participant from the study.
  The escalating X82 oral dose regimens were 50 mg alternate days, 50 mg daily, 100 mg alternate days, 100mg daily, 200mg daily, and 300mg daily.
Arm/Group | Dose Escalation of X-82 and Ranibizumab Rescue
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 3/35
Other Adverse Events (participants affected / at risk) | 28/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation of X-82 and Ranibizumab Rescue (N=35)
Chest pain (Cardiac disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 1 (1)
multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation of X-82 and Ranibizumab Rescue (N=35)
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Gastrointestinal reflux (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Urinary tract infection (Infections and infestations) | 5
Fatigue (General disorders) | 5
Sinusitis (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 2
Alanine amino transferase elevation (Hepatobiliary disorders) | 3
Aspartate amino transferase elevation (Hepatobiliary disorders) | 3
decrease body weight (General disorders) | 2
muscle spasma (Musculoskeletal and connective tissue disorders) | 3
arthritis (Musculoskeletal and connective tissue disorders) | 2
Headache (General disorders) | 4
Dizziness (General disorders) | 2
Dysgeusia (Gastrointestinal disorders) | 2
hypertension (Cardiac disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No